CLINICAL TRIAL: NCT03089463
Title: Foot Assessment in People With Diabetes: A Quantitative Diagnostic Approach
Status: Suspended | Type: Observational
Why Stopped: The study has not managed to recruit adequate number of participants.
Sponsor: Staffordshire University (Other)
Responsible Party: Principal Investigator, Roozbeh Naemi, Associate Professor of Biomechanics, Staffordshire University
Other Study IDs: 1
Record Dates: First submitted 2017-03-01; First posted 2017-03-24 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Diabetes; Diabetic Foot; Diabetes Complications; Diabetes; Neuropathic (Manifestation)
Keywords: Diabetes; Diabetic Foot; Biomechanics; Stratification; Diabetes Complications; Diabetes; Neuropathic (Manifestation); Risk Factors; Prospective Studies
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot; Diabetes Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation group: The entire participants in this study will be included in this group.
  Interventions: Diagnostic Test: Observation

INTERVENTIONS:
Diagnostic Test: Observation — The primary objective is to employ the measurements of neuropathy, micro/macro-perfusion, and biomechanics of the foot mainly tissue stiffness and plantar pressure to determine the vulnerability of foot to mechanical trauma and ulceration. From the data collected it is proposed that a prognostic risk stratification system will be developed based on the range of parameters collected to identify those that are at highest risk of ulceration incident. Those that are classed as high risk are to be sub-stratified to increase the accuracy of the system in predicting ulceration. This will allow a patient-specific approach to be taken in the prevention of ulcers by providing adequate information to predict ulceration incident.

SUMMARY:
This observational cohort study aims to develop a novel risk stratification system implementing biomechanics to aid in the prevention of diabetic foot ulcers.

DETAILED DESCRIPTION:
The purpose of this research observational cohort study is to investigate the applicability of using biomechanical assessment in predicting the ulceration incidence in patients with diabetic neuropathic feet. The proposed study will lead to the development of further stratification of high-risk patients into subcategories indicating the vulnerability of tissue to mechanical trauma, which deemed to be the leading cause of ulceration in people with diabetic neuropathy.

As it stands, the current systems used to evaluate the risk of diabetic foot rely on global parameters such as duration of diabetes and glycated hemoglobin to predict the likelihood and risk of diabetic foot ulceration. As ulceration happens as a result of repeat mechanical trauma to the foot that doesn't heal quickly enough due to other complications of diabetes, it is important to include mechanical measurements in predicting the ulceration incident in diabetic neuropathic patients. Despite this, the currently used risk stratification systems do not include biomechanics so by introducing biomechanics it will potentially be possible to predict the ulceration risk by using more local measurements.

The primary objective is to employ the measures of neuropathy, micro/macro-perfusion, and biomechanics of the foot mainly tissue stiffness and plantar pressure to determine the vulnerability of foot to mechanical trauma and ulceration. From the data collected it is proposed that a prognostic risk stratification system will be developed based on the range of parameters collected to identify those that are at highest risk of ulceration incident. Those that are classed as high risk are to be sub-stratified to increase the accuracy of the system in predicting ulceration. This will allow a patient-specific approach to be taken in the prevention of ulcers by providing adequate information to predict ulceration incident. This then can be used to determine the likelihood of an ulcer forming. Furthermore, the possibility of identifying the ulceration site will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 OR 2 diabetes
* Over 18
* English speaking
* Ability to walk unaided over 5m
* Diabetic neuropathy as defined by a 10g monofilament test

Exclusion Criteria:

* Lower limb surgery (amputation)
* Active ulcers
* History of neurological disorders (apart from neuropathy)
* Orthopaedic problems
* Systemic disease affecting mobility or leading to chronic inflammation of any lower limb joint.
* Visual impairment leading to difficulties in walking
* Charcot foot
* Unable to walk unaided for 5m

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants for this study will be recruited from the diabetic population of Staffordshire and Stoke-on-Trent Partnership and University Hospital North Midlands.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Qualitative foot assessment | April 2017 to April 2018 every 6 weeks
  The qualitative assessment is performed to identify if the patient has any foot or Nail fungi, and major foot deformities. Information regarding the toe deformities like clawed toes, hammer toe will also be recorded.
Skin assessment of the foot | April 2017 to April 2018 every 6 weeks
  This will be done when the patient lay down on their back on the couch with their bottom of the feet exposed where the measurements will be conducted. Photos will be taken from the plantar surface of the foot. This photos will be used in image processing software to identify any callus, foot and nail fungi and possible ulcers and their size.
Monofilament test | April 2017 to April 2018 every 6 weeks
  The next stage of tests will involve testing for signs of neuropathy, which is a loss of sensation in the foot caused by diabetes. To do this the three individual methods outline previously in the scientific background will be used. The 10g monofilament, which is a pen shaped device, which has a single filament similar to that of fishing line. The tip of the filament will be lightly pressed against nine key areas, big toes, middle toes, 1st metatarsal head, 3rd metatarsal head, 5th metatarsal head, left side of the mid foot, right side of the mid-foot, heel pad and the top surface of the foot. If there is a positive reaction then the next site can be examined if the test is negative then the site will be retested to decrease the possibility of error. If the outcome is negative again then it will be noted that they have lost sensation in that region of the foot. This will be done when the patient lay down on their back on the couch with their bottom of the feet exposed.
Tuning fork vibration test | April 2017 to April 2018 every 6 weeks
  Next the participant's sense of vibration will be measured using a 128Hz tuning fork. To do this the tuning fork is struck hard enough so that the vibration lasts roughly 30-40 seconds where it will be placed on either their sternum or wrist to get familiarised with the sensation of the vibration. Re-striking the tuning fork every time it will be placed on the top surface of the big toe, top surface of the midfoot and malleolus and with their eyes closed, the participant will be asked if they can feel the vibration and when it stops and the results will be recorded.This will be done when the patient lay down on their back on the couch with their bottom of the feet exposed where the measurements will be conducted.
Biothesiometry | April 2017 to April 2018 every 6 weeks
  The final part in checking for neuropathy is biothesiometery or measurement of vibration perception threshold (VPT). This involves a probe that vibrates at different amplitudes based on the amount of voltage supplied, normally up to 50V. As with the other tests the probe will be set to a high voltage setting and placed against the participant's wrist to feel the vibration before moving to their feet. The sites used are very similar to the monofilament test. The vibration will start at a low voltage setting and will slowly be increased until the participant can feel the vibration. Once they feel the vibration, the vibration will be stopped and the participant will be asked if they have noticed that it has stopped. This is to check that they do indeed have sensation in that area. If the voltage reaches 25V and no vibration is felt it can be deemed that the participant has lost sensation in that region.
Ankle Brachial Index | April 2017 to April 2018 every 6 weeks
  The next stage is to perform an ankle brachial index (ABI) test to determine if the participant has peripheral arterial dieses. ABI is the ratio between the highest systolic pressure at the ankle and the systolic pressure in arms. This is a common complication of diabetes where the blood vessels in the legs narrow or become completely blocked and as such, the blood flow to the legs decreases. To perform the test the participant will be asked to lie down on the couch and relax for about five minutes after that a blood pressure cuff is applied to the upper arm and a Doppler ultrasound is applied to the brachial artery and the blood pressure cuff is inflated until the blood flow can no longer be heard. At which point the blood pressure cuff will slowly be released until the flow can be heard again. The highest systolic pressure will be used to calculate ABI. For the ankle the blood pressure cuff is placed on the lower half of the shin and the same procedure is followed.
Transcutaneous oxygen pressure (TcPO2) | April 2017 to April 2018 every 6 weeks
  A TcPO2 test will also be performed, as this is another form of testing for problems with the circulation in the foot. This is performed with a probe that is heated to 44 degrees Celsius, which causes the blood vessels in the foot to expand, and induces local hyperthermia causing oxygen to pass through the skin towards a cathode. The test will be performed on the common locations for the probe are on the top of the foot, anteromedial calf approximately 10 cm below the knee and the thigh approximately 10cm above the knee. This will be done when the patient lay down on their back on the couch with their bottom of the feet exposed where the measurements will be conducted.
Skin Perfusion Pressure (SPP) | April 2017 to April 2018 every 6 weeks
  Another method that may be implemented in measuring the perfusion rate in the foot is that of skin perfusion pressure (SPP) this works by using a pressure cuff and a laser Doppler probe to establish hyperaemia in the area and measures the pressure that the blood returns to the capillaries following a controlled release. To do this a laser Doppler will be placed on the bottom surface of the foot and a pressure cuff will be placed over it. The cuff will then be inflated to 5 mm Hg initially and then the cuff is inflated to 20 mm Hg above the participants' brachial systolic pressure. The cuff is then deflated in 10 mm Hg steps every 5 seconds to a pressure of 50 mm Hg. The cuff is then deflated in 5 mm Hg steps every 15 seconds until the laser Doppler output increases for two consecutive pressure values. The pressure at which this first occurs is considered to be the SPP. This will be done when the patient lay down on their back on the couch.
Ankle/foot strength - Dynamometer | April 2017 to April 2018 every 6 weeks
  For measuring the ankle and foot strength a handheld dynamometer will be used, which measures the peak amount of force that is produced over a movement.
  To measure the muscle strength of the dorsiflexion movement the participant will be lying down on their back the participant with their knee held still by the researcher. This is to prevent additional movement and the recruitment of other muscles groups that could influence the results. With the knee now secured the handheld dynamometer is placed across the base of the toes (metatarsal heads) and the participant will be asked to pull their toes up towards themselves as hard as they can for five seconds with one minute rest in between each measurement. This will be repeated three times per foot. The same procedure will be employed for measuring the plantar flexion with the participant pushing their foot as hard as they can into the dynamometer. Again, the same procedure will be followed for testing inversion and eversion.
Range of motion (ROM) | April 2017 to April 2018 every 6 weeks
  To measure the ROM of the ankle a standard goniometer will be used where the participant will be asked to sit up onto the edge of the bed and dangle their feet. For dorsi/plantar flexion the fixed end of the goniometer will be placed on the bony prominence (lateral malleolus) pointing up the shin (fibula) and the participant will be asked to raise or lower their foot as far as they can. The free arm of the goniometer is then moved so that it is parallel with the bottom of the foot (5th metatarsal) and a reading is then taken.
  Furthermore a webcam perpendicular to the plane of motion will be used to take images of the foot during maximum plantar and dorsi flexion. The foot will be marked with a skin-friendly pen marker at anatomical landmarks on the medial and lateral side of the foot. This is to facilitate measuring the intersegmental foot range of motion as well as the ankle range of motion during dorsi and plantar flexion.
Foot Posture Index (FPI) | April 2017 to April 2018 every 6 weeks
  The participant will be asked to stand so that a foot posture index (FPI) test can be conducted. This is a test, which gives information as to how supinated or pronated the foot is. In simple terms this identifies if a person walks more on the inside of their foot or on the outside. The importance of this test is that it helps identifying the potential areas that are overloaded underneath the foot, and will provide valuable information. To perform a FPI the participant is asked to stand with both feet straight and parallel and the procedure according to Redmond 1998 will be followed.
Range of motion during walking | April 2017 to April 2018 every 6 weeks
  Before the plantar pressure test is performed, a number of anatomical landmarks will be marked on the participant's skin using skin-friendly markers. The markers will be placed on the lower extremity i.e. on the leg and the foot. During the test, a video camera will be set up at right angles to the pressure mat to record the gait of the participant. The recordings will be digitised to track the markers. From these measurements the ankle ROM during gait will be quantified.
Balance | April 2017 to April 2018 every 6 weeks
  The final test to be conducted is a balance test in which the participant will be asked to stand on the pressure mat with feet shoulder width apart and asked to try and keep their weight in the centre for thirty second and a recording will be taken and repeated three times. They will then close their eyes and repeat the same procedure that was followed for open eyes condition.
Gait Analyses | April 2017 to April 2018 every 6 weeks
  In addition to the measurements that are taken in the clinical setting some participants may be asked to participate in gait analyses and in shoe plantar pressure measurements. This would involve a separate session in the Biomechanics Lab at Staffordshire University. As part of the test the participant will be asked to have reflective markers attached to the skin and to walk over a force plate to measure the ground reaction forces and kinematics during movement.
Ultrasound elastography assessment | April 2017 to April 2018 every 6 weeks
  Ultrasound elastography allows an assessment of the stiffness of the plantar soft tissues at five different sites of the foot, 1st 3rd and 5th sub-metatarsal area, midfoot and Hallux. To conduct the test an interface material (ultrasound standoff) will be placed between the probe and the skin. This will add cushioning at the interface to prevent the applied force to the probe causing any damage to the foot. By applying minimal compression to the soft tissue through the compliant standoff a series of ultrasound images will be taken. These images will then be used with either elastography to look at plantar soft tissue stiffness.This will be done when the patient lay down on their back on the couch with their bottom of the feet exposed where the measurements will be conducted.
Blood test | April 2017 to April 2018 every 6 weeks
  The biochemistry of the participant's blood is also of great importance in the prediction as well as prevention of foot ulcers. These shall be collected with the participants consent from the central database. The parameters of interest are fasting blood sugar, PPBS, cholesterol, triglycerides, LDL, VLDL and HbA1c .
Thermography | April 2017 to April 2018 every 6 weeks
  A laser thermometer will be used to assess the locations on the foot that have previously experienced ulcers to look for a temperature difference. If the participant has not experienced a previous ulcer then the 1st, 3rd and 5th metatarsal heads, ball of the foot and the heel pad shall be examined for temperature changes.This will be done when the patient lay down on their back on the couch with their bottom of the feet exposed where the measurements will be conducted.
Barefoot Plantar pressure | April 2017 to April 2018 every 6 weeks
  One of the most important measures in this testing protocol is the measurement of plantar pressure. With the pressure mat calibrated the participant will be asked to walk over the mat six times three for the left foot and three for the right. This will allow an average pressure map for each foot to be calculated.
In-shoe plantar pressure measurement | April 2017 to April 2018 every 6 weeks
  The participants will also have a pressure sensitive insole placed within their shoe to study the pressure distribution during gait.
Perfusion measurement | April 2017 to April 2018 every 6 weeks
  Laser speckle contrast analysis technology will be utilised to study the blood flow on the plantar aspect of the foot. This will be done when the patient lay down on their back on the couch with their bottom of the feet exposed where the measurements will be conducted.

SECONDARY OUTCOMES:
Ulceration incident | April 2017 to April 2018 every 6 weeks
  Any ulceration incident and the site of ulceration will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Roozbeh Naemi, PhD, Principal Investigator — Staffordshire University; Nachiappan Chockalingam, Study Chair — Staffordshire University
Locations (1):
- Staffordshire University, Stoke-on-Trent, Staffordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No